CLINICAL TRIAL: NCT02519725
Title: ICU Diaries Impact of an ICU Diary on the Psychological Well-being of the Patients and Their Relatives. Mixed Multicenter Randomized Study With Blind Evaluation
Brief Title: Impact of an ICU Diary on the Well-being of Patients and Families. A Prospective Multicenter Mixed Study
Acronym: ICU-diary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Fondation de France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ICU DIARY
Record Dates: First submitted 2015-07-13; First posted 2015-08-11 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2016-06

CONDITIONS: Stress Disorders Post Traumatic
Keywords: Family; PTSD; Anxiety disorders; Depression disorders; Qualitative research
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the psychologist is blind for the study for assessing outcome measures
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With diary (Active Comparator): a ICU diary is open by staff for the patient and his relatives during the ICU stay
  Interventions: Other: ICU diary
- Without diary (No Intervention): No diary is open during the ICU stay

INTERVENTIONS:
Other: ICU diary — The intervention is the elaboration of an ICU diary by caregivers and families The first pages of the diary is standardized to include an explanation of the purpose of the diary. The diary is maintained by the family and ICU staff. The only instruction given to the families and staff members about diary entries is to refrain from writing about confidential matters that could not be shared among the patients, the staff and the relatives. Staff members are free to express compassion and their hope, or absence thereof, that the patient would recover. Relatives can speak freely with the patients without receiving guidance from the ICU staff. At the minimum, the ICU staff write a brief entry at each weekly staff meeting. For patients discharged to wards and if he can receive the diary, the diary is given to the patient. If the patient died, the diary is given to the family.
  Arms: With diary

SUMMARY:
The purpose of this study is to assess the influence of an ICU diary implemented during the ICU stay on the psychological well-being of patients and families after ICU discharge.

DETAILED DESCRIPTION:
Implementation of an ICU diary in a randomized design in 36 ICUs in France The ICU diary contains entries from staff and families or relatives

Quantitative description of psychological well-being of the patients and families or relatives are evaluated 3 months after ICU discharge

Qualitative evaluation of how the patient uses the diary is scheduled by a phone interview 6 months after ICU discharge.

An amendment of the ethic committee permitted to increase in 2016/02 both the number of eligible patients to 700 and the number of centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with his family admitted in an ICU and mechanically ventilated more than 48 hours

Exclusion Criteria:

* Patients without families admitted in an ICU and mechanically ventilated more than 48 hours
* Patients or families not fluent in French
* Patients moribund
* Patients with a neurologic or psychiatric disease responsible for admission or pre-existing before the ICU admission
* Patients admitted after a cardiac arrest
* Deaf and mute patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 715 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-08-09 (Actual)

PRIMARY OUTCOMES:
Post traumatic stress disorder symptoms in patients | 3 months after ICU discharge as measured by the Impact Evaluation Scale-Revised questionaire
  IES-R score > 22

SECONDARY OUTCOMES:
Post traumatic stress disorder symptoms in families | 3 months after ICU discharge as measured by the Impact Evaluation Scale-Revised questionaire
  IES-R score > 22
Anxiety and depression related symptoms in patients | 3 months after ICU discharge as measured by the Hospital Anxiety and Depression Scale
  HADS score > 8
Anxiety and depression related symptoms in families | 3 months after ICU discharge as measured by the Hospital Anxiety and Depression Scale
  HADS score > 8
Recollection of the memories of the ICU stay by the patient | 3 months after ICU discharge as measured by the memory tool questionnaire
  questionnaire ICU tool

OTHER OUTCOMES:
Use of the diary by the patient | 6 months after ICU discharge
  Qualitative research using phenomenology interpretative analysis and thematic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Maité Garrouste-Orgeas, MD, Principal Investigator — GHPSJoseph
Locations (1):
- Medical and surgical Intensive Care unit, Paris, France

REFERENCES:
- [Derived] Flahault C, Vioulac C, Fasse L, Bailly S, Timsit JF, Garrouste-Orgeas M. "A story with gaps": An interpretative phenomenological analysis of ICU survivors' experience. PLoS One. 2022 Mar 3;17(3):e0264310. doi: 10.1371/journal.pone.0264310. eCollection 2022. PMID 35239692
- [Derived] Garrouste-Orgeas M, Flahault C, Vinatier I, Rigaud JP, Thieulot-Rolin N, Mercier E, Rouget A, Grand H, Lesieur O, Tamion F, Hamidfar R, Renault A, Parmentier-Decrucq E, Monseau Y, Argaud L, Bretonniere C, Lautrette A, Badie J, Boulet E, Floccard B, Forceville X, Kipnis E, Soufir L, Valade S, Bige N, Gaffinel A, Hamzaoui O, Simon G, Thirion M, Bouadma L, Large A, Mira JP, Amdjar-Badidi N, Jourdain M, Jost PH, Maxime V, Santoli F, Ruckly S, Vioulac C, Leborgne MA, Bellalou L, Fasse L, Misset B, Bailly S, Timsit JF. Effect of an ICU Diary on Posttraumatic Stress Disorder Symptoms Among Patients Receiving Mechanical Ventilation: A Randomized Clinical Trial. JAMA. 2019 Jul 16;322(3):229-239. doi: 10.1001/jama.2019.9058. PMID 31310299
- [Derived] Garrouste-Orgeas M, Flahault C, Fasse L, Ruckly S, Amdjar-Badidi N, Argaud L, Badie J, Bazire A, Bige N, Boulet E, Bouadma L, Bretonniere C, Floccard B, Gaffinel A, de Forceville X, Grand H, Halidfar R, Hamzaoui O, Jourdain M, Jost PH, Kipnis E, Large A, Lautrette A, Lesieur O, Maxime V, Mercier E, Mira JP, Monseau Y, Parmentier-Decrucq E, Rigaud JP, Rouget A, Santoli F, Simon G, Tamion F, Thieulot-Rolin N, Thirion M, Valade S, Vinatier I, Vioulac C, Bailly S, Timsit JF. The ICU-Diary study: prospective, multicenter comparative study of the impact of an ICU diary on the wellbeing of patients and families in French ICUs. Trials. 2017 Nov 15;18(1):542. doi: 10.1186/s13063-017-2283-y. PMID 29141694
- See also: Impact of an intensive care unit diary on psychological distress in patients and relatives — http://www.ncbi.nlm.nih.gov/pubmed/22584757
- See also: Phenomenologic analysis of healthcare worker perceptions of intensive care unit diaries. — http://www.ncbi.nlm.nih.gov/pubmed/23336394
- See also: Writing in and reading ICU diaries: qualitative study of families' experience in the ICU. — http://www.ncbi.nlm.nih.gov/pubmed/25329581